CLINICAL TRIAL: NCT04724915
Title: Evaluation of Robot-assisted Total Knee Arthroplasty with Automatic Balancing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/1281bis
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Arm 1: Robot-assisted total knee arthroplasty Arm 2: Conventional jig-based total knee arthroplasty
Who Masked: Outcomes Assessor
Masking Description: Masked investigators will be responsible for the data processing and analysis. Reporting will be done together with non-masked authors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robot-assisted TKA (Experimental): Patients undergoing TKA with the assistance of robot technology.
  Interventions: Procedure: Robot-Assisted Total Knee Arthroplasty
- Conventional TKA (Active Comparator): Patients undergoing TKA with manual instrumentarium
  Interventions: Procedure: Conventional Total Knee Arthroplasty

INTERVENTIONS:
Procedure: Conventional Total Knee Arthroplasty — People will undergo surgery to replace the knee joint with a prosthesis in case of osteoarthritis. This will be performed with manual instrumentarium (jig-based).
  Arms: Conventional TKA
Procedure: Robot-Assisted Total Knee Arthroplasty — People will undergo surgery to replace the knee joint with a prosthesis in case of osteoarthritis. This will be performed with the help of a surgical robot.
  Arms: Robot-assisted TKA

SUMMARY:
The goal is to evaluate the outcomes and learning curve of a robot-assisted total knee arthroplasty device with automatic ligament balancing.

ELIGIBILITY:
Inclusion Criteria:

* End stage osteoarthritis of the knee joint with failed conservative treatment

Exclusion Criteria:

* Previous ligament trauma of the MCL/LCL
* Previous fracture of femur or tibia
* Fixed flexion contracture > 10°
* Flexion < 110°
* Coronal deformity > 15°
* Previous infection of the knee joint
* Ligament insufficiency
* Neurologic conditions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Knee Laxity | Preoperative and postoperatively at 1 year.
  Coronal knee laxity will be evaluated with stress examination. Coronal stress will be evaluated with a stress radiograph. The deviation between the neutral position and position under stress will be measured on a coronal radiograph. The angle between the joint lines will be measured on the coronal radiograph.

SECONDARY OUTCOMES:
Patient reported outcome measures | Preoperative
  The following patient reported outcome measures will be evaluated: Knee Injury and Osteoarthritis outcome score. The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems
Patient reported outcome measures | Preoperative
  The following patient reported outcome measures will be evaluated: Knee Society Score. The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
Patient reported outcome measures | Preoperative
  The following patient reported outcome measures will be evaluated: EuroQoL. The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
Patient reported outcome measures | Preoperative
  The following patient reported outcome measures will be evaluated: Pain Catastrophizing Scale. The score is a percentage score from 0 to 52, 0 representing no problems and 52 representing extreme problems.
Change in patient reported outcome measures | Postoperatively at 6 weeks, 6 months, 1 year and 2 years.
  The change for the following patient reported outcome measures will be evaluated (compared to preoperatively): Forgotten Joint Score. The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
Change in patient reported outcome measures | Postoperatively at 6 weeks, 6 months, 1 year and 2 years.
  The change for the following patient reported outcome measures will be evaluated (compared to preoperatively): Knee Injury and Osteoarthritis outcome score. The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
Change in patient reported outcome measures | Postoperatively at 6 weeks, 6 months, 1 year and 2 years.
  The change for the following patient reported outcome measures will be evaluated (compared to preoperatively): Knee Society Score. The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
Change in patient reported outcome measures | Postoperatively at 6 weeks, 6 months, 1 year and 2 years.
  The change for the following patient reported outcome measures will be evaluated (compared to preoperatively): EuroQoL. The score is a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
Change in patient reported outcome measures | Postoperatively at 6 weeks, 6 months, 1 year and 2 years.
  The change for the following patient reported outcome measures will be evaluated (compared to preoperatively): Pain Catastrophizing Scale. The score is a percentage score from 0 to 52, 0 representing no problems and 100 representing extreme problems.
Alignment | Preoperative and postoperatively at 6 weeks and 6 months.
  Coronal alignment on xrays. The lateral distal femoral angle (LDFA) will be evaluated. This is the angle between the mechanical femoral axis and the line between the distal articular surface of the femur. Additionally the medial proximal tibial angle (MPTA) will be evaluated. This is the line between the condylar surface and the mechanical axis of the tibia on a coronal radiograph.
Knee laxity anteroposterior | Preoperative and postoperatively at 1 year.
  Sagittal knee laxity will be evaluated with stress examination. Sagittal knee laxity will be measured with an anteroposterior laxitymeter (GENOUROB; CE Marked). With a standardized setup, anteroposterior laxity can be obtained by measuring the anteroposterior deviation from the neutral position with up to 300 Newton of force.
Knee kinematics in 3D after squat, knee flexion/extension, stair ascend and descend. | Postoperatively at 1 year.
  Knee kinematics in 3D obtained with fluoroscopy. Patients will be asked to perform squats, a flexion/extension movement, ascend and descend stairs. 3D motion of the prosthesis components can be obtained by projecting the 3D file of the prosthesis components onto the fluoroscopy images.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Victor, MD, PhD, Study Chair — UZ Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vermue H, Arnout N, Tampere T, Stroobant L, Dereu A, Victor J. Standardized Intraoperative Robotic Laxity Assessment in TKA Leads to No Clinically Important Improvements at 2 Years Postoperatively: A Randomized Controlled Trial. Clin Orthop Relat Res. 2025 Oct 1;483(10):1866-1874. doi: 10.1097/CORR.0000000000003505. Epub 2025 Apr 16. PMID 40258174